CLINICAL TRIAL: NCT03237195
Title: Utility and Cost-effectiveness of Microscopic Examination of the Neck Dissection Specimen in Its Entirety.
Brief Title: Utility and Cost-effectiveness of Microscopic Examination of the Neck Dissection.
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-0288
Record Dates: First submitted 2017-07-28; First posted 2017-08-02 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2017-07

CONDITIONS: Metastasis
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Neck Dissection

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: additional soft tissue in neck dissections — Evaluation of submission of additional soft tissue in neck dissections for head and neck squamous cell carcinomas

SUMMARY:
Most patients with cancer of the head and neck are offered surgical resection of the primary tumor. In order to determine how the tumor will eventually behave, along with the resection of the primary tumor, lymph nodes present in the neck are also dissected. Different institutes have different protocol on handling of the specimen that is received by the pathology labs after dissection of the neck. The investigators intend to analyze the protocol that they use to evaluate the neck dissection specimen.

DETAILED DESCRIPTION:
This will be a retrospective study. All neck dissections received in the histology laboratory from Jan 2013 to December 2016 will be retrieved from the histopathology files by conducting a search through CoPath. The glass slides of all the neck dissections that fit the study criterion will be retrieved from the archives. The glass slides will be reviewed by the pathologist.

At the time of review number of lymph nodes identified microscopically, presence or absence of metastasis and if the Lymph Nodes (LN) were palpable or not palpable will be documented. The data will be analyzed to see if the submission of extra fat yielded any additional positive lymph nodes or microscopic deposits. The cost analysis for additional slides will be also done.

ELIGIBILITY:
Inclusion Criteria:

1. Neck dissection (unilateral and/or bilateral)
2. Primary squamous cell carcinoma of head and neck

Exclusion Criteria:

1. Any neck dissection performed outside UMMC and case received as a consult.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent neck dissection for squamous cell carcinomas of head and neck origin.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of additional lymph nodes obtained with additional sampling of soft tissue | 3 years
  Number of additional lymph nodes obtained with additional sampling of soft tissue

CONTACTS AND LOCATIONS:
Overall Officials: Varsha Manucha, Principal Investigator — Associate Professor
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gillies EM, Luna MA. Histologic evaluation of neck dissection specimens. Otolaryngol Clin North Am. 1998 Oct;31(5):759-71. doi: 10.1016/s0030-6665(05)70085-2. PMID 9735105
- [Result] Jose J, Coatesworth AP, MacLennan K. Cervical metastases in upper aerodigestive tract squamous cell carcinoma: histopathologic analysis and reporting. Head Neck. 2003 Mar;25(3):194-7. doi: 10.1002/hed.10194. PMID 12599286
- [Result] Seethala RR. Current state of neck dissection in the United States. Head Neck Pathol. 2009 Sep;3(3):238-45. doi: 10.1007/s12105-009-0129-y. Epub 2009 Aug 7. PMID 20596978
- [Result] Muirhead D, Aoun P, Powell M, Juncker F, Mollerup J. Pathology economic model tool: a novel approach to workflow and budget cost analysis in an anatomic pathology laboratory. Arch Pathol Lab Med. 2010 Aug;134(8):1164-9. doi: 10.5858/2000-0401-OA.1. PMID 20670137
- [Result] van den Brekel MW, Stel HV, van der Valk P, van der Waal I, Meyer CJ, Snow GB. Micrometastases from squamous cell carcinoma in neck dissection specimens. Eur Arch Otorhinolaryngol. 1992;249(6):349-53. doi: 10.1007/BF00179388. PMID 1384570